CLINICAL TRIAL: NCT04335084
Title: A Randomized, Double-Blind, Placebo-Controlled Phase IIa Study of Hydroxychloroquine, Vitamin C, Vitamin D, and Zinc for the Prevention of COVID-19 Infection
Brief Title: A Study of Hydroxychloroquine, Vitamin C, Vitamin D, and Zinc for the Prevention of COVID-19 Infection
Acronym: HELPCOVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Collaborators: DSCS CRO (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: PRG-042
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: COVID-19; Coronavirus Infection; Sars-CoV2; Corona Virus Infection; COVID; Coronavirus; Coronavirus-19; Coronavirus 19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Hydroxychloroquine; Ascorbic Acid; Vitamin D; Zinc

STUDY DESIGN:
Intervention Model Description: This study will focus on medical workers who at elevated risk of COVID-19 due to exposure to positive patients in the Emergency Department or Intensive Care Unit
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Medical Workers (Experimental): Medical workers who are exposed to COVID-19 and as such are at higher risk for infection.
  Interventions: Drug: Hydroxychloroquine; Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin D; Dietary Supplement: Zinc
- Placebo (Placebo Comparator): Medical workers who are exposed to COVID-19 and as such are at a higher risk for infection
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin D; Dietary Supplement: Zinc

INTERVENTIONS:
Drug: Hydroxychloroquine — Prophylaxis treatment for COVID-19
  Other Names: Plaquenil
  Arms: Medical Workers
Dietary Supplement: Vitamin C — Prophylaxis treatment for COVID-19
Dietary Supplement: Vitamin D — Prophylaxis treatment for COVID-19
Dietary Supplement: Zinc — Prophylaxis treatment for COVID-19

SUMMARY:
This is a Phase II interventional study testing whether treatment with hydroxychloroquine, Vitamin C, Vitamin D, and Zinc can prevent symptoms of COVID-19

DETAILED DESCRIPTION:
In this study, subjects will take a regimen of hydroxychloroquine, vitamin C, vitamin D, and Zinc to test if this combination can prevent COVID-19. Treatment with hydroxychlorquine will last 1 day. Treatment with vitamin C, vitamin D, and and zinc will last 12 weeks. The study will last 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent, provided electronically via the EDC, demonstrating the subject understands the procedures required for the study and the purpose of the study
2. Male or female patients 18 years of age or older that are considered to be high-risk individuals.

   a. High-risk individuals are defined as all health care workers in hospitals, clinics, and emergency rooms, and medical facilities.
3. Subjects must agree to practice at least two highly effective methods of birth control for the duration of the study This includes condoms with spermicide, oral birth control pills, contraceptive implants, intra-uterine devices, or diaphragms. At least one of these must be a barrier method. Subjects not of reproductive potential will be exempt (e.g. post-menopausal, surgically sterilized)

Exclusion Criteria:

1. Refusal to provide informed consent
2. Any previous positive test for COVID-19 by RT-PCR
3. Symptomatic for COVID-19
4. Diarrhea prior to the start of treatment
5. Type I or II diabetes
6. Atherosclerotic Coronary Artery Disease
7. Any contraindication for treatment with hydroxychloroquine including:

   1. Hypoglycemia
   2. G6PD deficiency
   3. Porphyria
   4. Anemia
   5. Neutropenia
   6. Alcoholism
   7. Myasthenia Gravis
   8. Skeletal muscle disorder
   9. Maculopathy
   10. Changes in the visual field
   11. Liver disease, with ALT/AST > 2.5 upper limit normal and total bilirubin >2.5 upper limit normal
   12. Psoriasis
   13. Any contraindicated medications found in Appendix 2
8. Any comorbidities which, in the opinion of the investigator, constitute health risk for the subject.
9. Vaccination for SARS-CoV-2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2024-04-11 (Actual)

PRIMARY OUTCOMES:
Prevention of COVID-19 symptoms as recorded in a daily diary | 24 weeks
  Any symptoms of COVID-19 will be recorded in a daily diary. Symptoms (including fever measured in degrees Fahrenheit, dry cough, productive cough, difficulty speaking, wheezing, dry mouth, headache, chest tightness, difficulty with exertion, shortness of breath, sore throat, malaise, and diarrhea) will be rated as not present, mild, moderate, or severe.
Safety as determined by presence or absence of Adverse Events and Serious Adverse Events | 24 weeks
  To assess the presence or absence of side effects (graded 1-5), and whether they are tolerable (grade 1-2). AE and SAE will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banjanac M, Munic Kos V, Nujic K, Vrancic M, Belamaric D, Crnkovic S, Hlevnjak M, Erakovic Haber V. Anti-inflammatory mechanism of action of azithromycin in LPS-stimulated J774A.1 cells. Pharmacol Res. 2012 Oct;66(4):357-62. doi: 10.1016/j.phrs.2012.06.011. Epub 2012 Jul 3. PMID 22766077
- [Background] Cortegiani A, Ingoglia G, Ippolito M, Giarratano A, Einav S. A systematic review on the efficacy and safety of chloroquine for the treatment of COVID-19. J Crit Care. 2020 Jun;57:279-283. doi: 10.1016/j.jcrc.2020.03.005. Epub 2020 Mar 10. PMID 32173110
- [Background] Gao J, Tian Z, Yang X. Breakthrough: Chloroquine phosphate has shown apparent efficacy in treatment of COVID-19 associated pneumonia in clinical studies. Biosci Trends. 2020 Mar 16;14(1):72-73. doi: 10.5582/bst.2020.01047. Epub 2020 Feb 19. PMID 32074550
- [Background] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Background] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466